CLINICAL TRIAL: NCT04730518
Title: Yoga-based Group Intervention for In-Patients With Schizophrenia Spectrum Disorder - a Rater-Blinded Randomized Controlled Trial
Brief Title: Yoga-based Group Intervention (YoGI) for In-patients With Schizophrenia Spectrum Disorders
Acronym: YING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Kerem Böge, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YING2021
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: A rater-blinded randomized controlled trial with a parallel group design is used. The participants in the control group receive the usual treatment (TAU), while the experimental group receives yoga-based group intervention (YoGI) in addition to TAU.
Who Masked: Outcomes Assessor
Masking Description: A blinded psychologist or psychiatrist who works independently of the (co-) psychologist conducts the rater-questionnaires. Due to the psychotherapeutic nature of the study, information about the treatment allocation has to be shared with the co-psychologist and the participants. Randomization is conducted by the Random Group Generator (pubmed, 2018).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga-based Group Intervention (YoGI) (Experimental): The yoga-based group intervention (YoGI) involves a four-week intervention with weekly group therapy sessions in addition to TAU. The fifty-minute session takes place with a group size of max. 10 participants and was held once a week by a psychologist who is also a trained yoga-teacher.
  A yoga session starts with breathing exercises (pranayama), followed by various exercises in standing, sitting and lying down (asanas), which are accompanied by mindful instructions from the psychologist. Every yoga session ends with a final relaxation (shavasana), which can take the form of a body scan, for example.
  Interventions: Behavioral: Yoga-based group intervention (YoGI)
- Treatment as usual (TAU) (Active Comparator): Treatment as usual (TAU) at the ward consists of a variety of daily group therapies the patients partake in. Every patient at the ward receives a daily schedule depending on individual needs for therapy. The therapies offered at the ward include occupational therapy, physiotherapy, psychoeducative groups, and concentration practice of two levels, all not related to mindfulness interventions. In addition to the group activities at the ward, every patient receives individual psychotherapy sessions (CBTp) at least once a week, held by a certified psychiatrist or psychologist. Psychopharmacological treatment is provided by the physicians, and social workers are available in order to support patients in managing their everyday lives after the stationary treatment. Weekly group meetings at the ward, together with the treating physicians, psychologists, psychotherapists, social workers and the respective patient, foster the exchange success and possible improvements of the treatment.
  Interventions: Behavioral: Yoga-based group intervention (YoGI)

INTERVENTIONS:
Behavioral: Yoga-based group intervention (YoGI) — see above

SUMMARY:
A rater-blinded randomized controlled trial with a parallel-group design is utilized, comprised of yoga-based group intervention (YoGI) in the experimental condition, and treatment as usual (TAU) in the control condition. The participants in the experimental condition participate in YoGI beside their regular psychiatric treatment (TAU). The intervention is designed for in-patients with schizophrenia spectrum disorders. With the aim of examining the feasibility, acceptability and effectiveness, self-report and blinded rater-based assessments are evaluated before the YoGI (T0), and after four weeks of taking part in intervention (T1).

Building on the results of the feasibility and acceptability trial, the study is now progressing to a full randomized controlled trial. The primary outcome for the full trial will be positive symptoms of schizophrenia spectrum disorders, assessed by a blinded rater using the Positive and Negative Syndrome Scale (PANSS). The target sample size has been adjusted to ensure sufficient statistical power, and the trial will evaluate secondary outcomes, including (body) mindfulness, negative symptoms, cognitive functioning, and quality of life, and stress. This study aims to provide robust evidence for the effectiveness of YoGI in comparison to treatment as usual (TAU).

DETAILED DESCRIPTION:
Psychiatrists and psychologists at the ward for psychotic disorders identify eligible participants and invite them to participate in the study. An eligibility screening is held by the study assistant at baseline, introducing the study, providing informed electronic consent, as well as conducting the self-report measures and app-based assessments. A blinded psychologist who works independently of the (co-) psychologist conducts the remaining rater-questionnaires. Due to the psychotherapeutic nature of the study, information about the treatment allocation had to be shared with the co-psychologist and the participants. Saliva samples are also taken to examine stress-related biomarkers. Randomization was conducted by the Random Group Generator (pubmed, 2018). The data management plan includes standard procedures for data-handling such as using anonymized identification codes for patient data. The participants have the right to access their data, and the right to claim an annihilation. The data is being saved in an online database, only allowing researchers involved in the study to access the data.

ELIGIBILITY:
Inclusion Criteria:

* male and female participants
* treated as psychiatric inpatients at the psychosis ward or in the social-psychiatric day clinic
* ≥18 years
* diagnosis of a schizophrenia-spectrum disorder according to the Diagnostical and Statistical Manual 5th edition) and the International Statistical Classification of Diseases and Related Health Problems(ICD-10) code F2
* ability to give informed consent
* willingness and ability to engage in psychotherapeutic group therapy
* low to moderate psychotic state indicated with a score of ≤ 6 for each item at the Positive scale of the Positive and Negative Syndrome Scale (PANSS, Peralta & Cuesta, 1994)

Exclusion Criteria:

* a score > 6, suggesting an acute psychotic episode with severe psychotic symptoms (Peralta& Cuesta, 1994)
* acute suicidality, assessed by item eight of the Calgary Depression Scale for Schizophrenia > 1 (Addington, Addington, Maticka-Tyndale, & Joyce, 1992)
* any neurological disorders that may affect cognitive functioning
* acute substance abuse other than nicotine and prescribed medication
* conflicting co-therapy such as electroconvulsive therapy or ketamine treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
PANSS Symptomatology - Positive and Negative Symptoms | 18 months
  Positive Symptoms as measure by the Positive and Negative Syndrome Scale (PANSS) to assess symptoms on a scale from 1 (non-existent) to 7 (extremely severe, 14 questions)
Proportion of pp receiving threshold dose (Acceptability) | 18 months
  The proportions of participants receiving a threshold dose of the intervention (50% or more) and the proportion of participants with outcome measures at post-intervention and data completion. (Adherence and retention rate)
Nr. of pp willing to participate in YoGI (Operational Feasibility) | 18 months
  The number of eligible participants that are willing to participate in YoGI (recruitment)

SECONDARY OUTCOMES:
SMQ Mindfulness | 18 months
  Southampton mindfulness questionnaire (SMQ), 16 items on a scale from 1 (applies fully) to 7 (does not apply at all)
BMQ Body Mindfulness | 18 months
  Body Mindfulness Questionnaire (BMQ), 14 items on a scale from 1 (not at all) to (5) every day
DASS Symptoms - Depression and Anxiety | 18 months
  Depression Anxiety Stress Scales (DASS), 21 questions that can be answered on a scale from 0 (does not apply to me) to 3 (applies to me strongly/most of the time)
PSP Personal and Social Performance | 18 months
  Personal and Social Performance Scale (PSP), Interview measures personal and social functioning in the domains of: Socially useful activities (eg, work and study), Personal and social relationships, Self-care, Disturbing and aggressive behaviors. Different domains are rated on a scale from absent to highly severe.
CFQ Cognitive Fusion | 18 months
  Cognitive Fusion Questionnaire (CFQ), 7 questions that can be answered on a scale from 1(not applicable) to 7 (applies always)
WHO-QOL-Bref Quality of Life - domains assessed include physical and psychological health, social relationships and environment | 18 months
  World Health Organisation Quality of Life (WHO-QOL-Bref) to assess quality of life measured on a scale from 1 (never) to 5 (always). Facets incorporated in the 4 domains: 1. Physical health - Activities of daily living Dependence on medicinal substances and medical aids Energy and fatigue Mobility Pain and discomfort Sleep and rest Work Capacity; 2. Psychological - Bodily image and appearance Negative feelings Positive feelings Self-esteem Spirituality / Religion / Personal beliefs Thinking, learning, memory and concentration; 3. Social relationships - Personal relationships Social support Sexual activity; 4. Environment - Financial resources Freedom, physical safety and security Health and social care: accessibility and quality Home environment Opportunities for acquiring new information and skills Participation in and opportunities for recreation / leisure activities Physical environment (pollution / noise / traffic / climate) Transport.
CANTAB Broad Cognitive Functioning | 18 months
  CANTAB mobile App to assess cognitive functioning, validated version for schizophrenia
SSTICS Subjective Cognitive Functioning | 18 months
  Subjective Scale to Investigate Cognition (SSTICS), 21 items from a scale from 1 to 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Universitätsmedizin Berlin, Campus Benjamin Franklin, Steglitz, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No